CLINICAL TRIAL: NCT00754364
Title: A Randomized Phase II Study of Progression Free Survival Comparing Gemcitabine (1000 mg/m2 Infusion) Versus Carboplatin (AUC5 Infusion) Plus Alimta (500 mg/m2 Infusion) as First-line Chemotherapy in Elderly Patients With Locally Advanced (Stage IIIb) or Metastatic (Stage IV) Non Small Cell Lung Cancer (NSCLC)
Brief Title: Mono Versus Polichemotherapy in Non Small Cell Lung Cancer (NSCLC) Elderly Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low enrollment rate
Sponsor: Armando Santoro, MD (Other)
Responsible Party: Sponsor-Investigator, Armando Santoro, MD, MD, Istituto Clinico Humanitas
Organization: Istituto Clinico Humanitas (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ONC-2007-003
Record Dates: First submitted 2008-09-17; First posted 2008-09-18 (Estimated); Last update posted 2022-09-10 (Actual); Status verified 2022-09

CONDITIONS: NSCLC
MeSH Terms: interventions — Pemetrexed; Carboplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pemetrexed/Carboplatin (Experimental): Pemetrexed (500 mg/m2 infusion) plus Carboplatin (AUC5 infusion)
  Interventions: Drug: Pemetrexed/Carboplatin
- Gemcitabine (Active Comparator): Gemcitabine 1250 mg/mq
  Interventions: Drug: Gemcitabine

INTERVENTIONS:
Drug: Pemetrexed/Carboplatin — Patients will receive Pemetrexed intravenous infusion (i.v.) via infusion pump or gravity drip, at a dose of 500 mg/m2 (over a target of 10 minutes). Pemetrexed should be administered every 21 days on the same day.
  Patients will receive carboplatin intravenous continuous infusion (i.v.) over 30 minutes via infusion pump or gravity drip, at a dose of AUC5. Carboplatin should be administered every 21 days on the same day.
  Arms: Pemetrexed/Carboplatin
Drug: Gemcitabine — Patients will receive gemcitabine 1250 mg/m2 as a 30 minutes intravenous infusion on days 1 and 8 and of a 21-day cycle.Patients may continue to receive gemcitabine for up to a maximum of 6 cycles.
  Arms: Gemcitabine

SUMMARY:
Between 10% and 25% of newly diagnosed stage IIIB/stage IV patients currently receive single agent chemotherapy regimens. A significant proportion of these patients will be elderly (70 years of age) and many oncologists would consider intravenous vinorelbine or gemcitabine to be the standard of care in this patient population. It has been demonstrated that single agent vinorelbine offers therapeutic advantages to selected NSCLC patients over best supportive care alone.

Carboplatin plus Alimta have an acceptable toxicity profile and few clinical problems so it could be acceptable its use in elderly patients.

A randomised study is being performed therefore to assess whether progression free survival, the primary efficacy endpoint for this study, achieved with Carboplatin plus Alimta is superior than achieved with gemcitabine, one of the current standards of care in elderly patients with advanced NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* NSCLC, locally advanced (stage IIIB) or metastatic (stage IV) disease, not amenable to curative surgery or radiotherapy
* Female or male patients aged 70 years and over
* Measurable disease according to RECIST criteria, with at least one measurable lesion
* No prior chemotherapy, biological or immunological therapy
* Adeguate hepatic, renal and bone marrow function
* ECOG Performance Status ≤ 2
* Life expectancy of at least 12 weeks

Exclusion Criteria:

* Newly diagnosed CNS metastases that have not been treated with surgery or radiation
* Less than 4 weeks since completion of prior radiotherapy or persistence of any radiotherapy related toxicity
* Any other experimental or anti-cancer therapy within 30 days before study drug administration
* Concurrent treatment with any other experimental or anti-cancer therapy

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 108 (Actual)
Dates: Start 2008-10; Primary Completion 2014-05 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Evaluate Progression Free Survival of Carboplatin plus Alimta vs gemcitabine in chemonaive, elderly stage IIIB-IV NSCLC patients. | Efficacy after the inclusion of the last patient

SECONDARY OUTCOMES:
Overall Survival Quality of life | After the follow up period

CONTACTS AND LOCATIONS:
Overall Officials: Armando Santoro, MD, Principal Investigator — Istituto Clinico Humanitas
Locations (1):
- Istituto Clinco Humanitas, Rozzano, Milan, Italy